CLINICAL TRIAL: NCT01955850
Title: Online or Face-to-face Treatment for Insomnia? A Wait-list Controlled Trial
Brief Title: Online or Face-to-face Treatment for Insomnia?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: Slaapmakend (Unknown)
Responsible Party: Principal Investigator, Jaap Lancee, PhD, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UvA-2013-KP-3125
Record Dates: First submitted 2013-09-20; First posted 2013-10-08 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

ARMS (3):
- Internet-delivered CBT for insomnia (Experimental): Online Cognitive behavioral treatment for insomnia
  Interventions: Behavioral: Cognitive behavioral treatment for insomnia
- Face-to-face CBT for insomnia (Experimental): Face-to-face Cognitive behavioral treatment for insomnia
  Interventions: Behavioral: Cognitive behavioral treatment for insomnia
- Waiting-list (No Intervention): Waiting-list

INTERVENTIONS:
Behavioral: Cognitive behavioral treatment for insomnia — Cognitive behavioral treatment for insomnia, consisting of: psycho-education, sleep hygiene, stimulus control, sleep restriction, cognitive therapy.
  Arms: Face-to-face CBT for insomnia; Internet-delivered CBT for insomnia

SUMMARY:
The object of this study is to compare internet-delivered treatment for insomnia to face-to-face treatment and a waiting-list. In this study participants are randomized to: 1) online cognitive-behavioral intervention; 2) face-to-face cognitive behavioral intervention; 3) waiting-list. Both the online and face-to-face interventions consist of: diary; psycho-education; relaxation exercises; stimulus control/sleep hygiene; sleep restriction; challenging the misconceptions about sleep; and paradoxical exercise. Adult persons with insomnia will be invited via a popular scientific website to fill out online questionnaires. Participants fill out questionnaires and a dairy at baseline post-test, 3-month follow-up, and 6-month follow-up. Participants on the waiting-list receive online treatment after the first post-test. The investigators expect that the online-delivered treatment and the face-to-face treatment are equally effective.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia disorder according to DSM-5
* Sleep onset latency/wake after sleep onset > 30 minutes , three times or more a week
* Insomnia three months or longer
* Access to internet
* Possibility to travel to one of the treatment sites

Exclusion Criteria:

* Earlier cognitive behavioral treatment for insomnia
* Start other psychological treatment in the last 6 months
* Doing shift work
* Major depression disorder
* Pregnancy or breast feeding
* Schizophrenia or psychosis
* Suicidal plans
* Sleep apnea
* drugs or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sleep continuity (consisting of sleep latency, time awake after sleep onset, total sleep time) | Change from baseline to post-test, 3-months, and 6-months follow-up
  For sleep continuity a 7-day sleep diary is used based on the consensus sleep diary.
Insomnia Severity Index | Change from baseline to post-test, 3-months, and 6-months follow-up

SECONDARY OUTCOMES:
Anxiety (HADS-A) | Change from baseline to post-test, 3-months, and 6-months follow-up
Sleep related worry measured with the Anxiety and Pre-occupation about Sleep Scale | Change from baseline to post-test, 3-months, and 6-months follow-up
Sleep related arousal measured with the Pre-arousal sleep scale | Change from baseline to post-test, 3-months, and 6-months follow-up
Sleep related cognitions measured with the Dysfunctional Beliefs and Attitudes about sleep scale (DBAS) | Change from baseline to post-test, 3-months, and 6-months follow-up
Sleep medication usage per day measured with the sleep diary | Change from baseline to post-test, 3-months, and 6-months follow-up
Depression measured with the CES-D | Change from baseline to post-test, 3-months, and 6-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Lancee, PhD, Principal Investigator — University of Amsterdam
Locations (1):
- Department of Clinical Psychology, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Lancee J, van den Bout J, van Straten A, Spoormaker VI. Internet-delivered or mailed self-help treatment for insomnia?: a randomized waiting-list controlled trial. Behav Res Ther. 2012 Jan;50(1):22-9. doi: 10.1016/j.brat.2011.09.012. Epub 2011 Oct 24. PMID 22055281
- [Derived] Lancee J, van Straten A, Morina N, Kaldo V, Kamphuis JH. Guided Online or Face-to-Face Cognitive Behavioral Treatment for Insomnia: A Randomized Wait-List Controlled Trial. Sleep. 2016 Jan 1;39(1):183-91. doi: 10.5665/sleep.5344. PMID 26414893
- See also: General website for insomnia and used for the recruitment — http://www.insomnie.nl